CLINICAL TRIAL: NCT05113706
Title: Does Bystanders Emotional State Influence Dispatcher-assisted Cardiopulmonary Resuscitation?
Brief Title: Does Bystanders Emotional State Influence Dispatcher-assisted Cardiopulmonary?Resuscitation
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Emergency Medical Services, Capital Region, Denmark (Other Government)
Responsible Party: Sponsor
Other Study IDs: F35150-04
Record Dates: First submitted 2021-10-28; First posted 2021-11-09 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-02

CONDITIONS: Out-Of-Hospital Cardiac Arrest; Emotional Distress
Keywords: Dispatcher; Emergency call; Out-Of-Hospital Cardiac Arrest
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bystander not emotional distressed: If caller is not emotional distressed the first minute of the call
- Bystander emotional distressed: If caller is emotional distressed the first minute of the call

SUMMARY:
The study aims to investigate bystanders' emotional stress state in out-of-hospital cardiac arrest (OHCA) emergency calls and the association with the quality of dispatcher-assisted cardiopulmonary resuscitation (DA-CPR).

DETAILED DESCRIPTION:
Delayed CPR is believed to be an important factor in the outcome of out-of-hospital cardiac arrest (OHCA). Bystanders' emotional stress state might affect recognition of cardiac arrest and the resuscitation attempt. The study aims to investigate the association between a bystander's emotional stress state at the beginning of the emergency call in out-of-hospital cardiac arrest (OHCA) and dispatcher-assisted cardiopulmonary resuscitation (DA-CPR).

Method

The study is a retrospective and observational study of OHCA emergency calls from the capital region of Denmark from 01.09.2018 - 01.11.2019. The audio recordings of the emergency calls will be obtained from the emergency medical service database. A code catalogue with standardised default descriptions to each variable will be used. The study will only include the first person whom the medical dispatcher talk to. The rating of the calls will be performed by five observers outside of the research group, who have no conflict of interest.

The primary outcome of the present study will be to investigate an association between a bystander's emotional stress state in the beginning of the emergency call of OHCA and the time until first chest compression. Secondarily, the study investigated the association between the bystander's emotional stress and:

Outcome variables:

1. Time to recognition of OHCA, time to initiate CPR, and time to first compression.
2. Assessment of OHCA by the medical dispatcher (Does the dispatcher address patient breathing status and consciousness) (Yes/No)
3. The quality of DA-CPR instructions:

   1. Was the medical dispatcher motivating and encouraging when giving instructions (Yes/No)
   2. Was the medical dispatcher assertive or passive when giving instructions (Yes/No)
   3. Did the medical dispatcher instruct on depth and speed of compressions (Yes/No) Information about caller such as gender and relationship to the patient will also be included in the analyse.

Descriptive analysis of baseline characteristics of emergency calls and dispatchers will be performed by frequency distributions (N %) stratified by emotional stress.

Investigators will use logistic regression on categorical variables to analyse differences in the quality of DA-CPR based on the emotional stress state.

Wilcoxon rank-sum test will be used on non-normally distributed continuous variables to analyse differences in time until first chest compression. Two-way ANOVA will be used to analyse the mean of quantitative variables according to the levels of categorical variables. Furthermore, failure analysis was used to analyse and visualise differences in time until chest compressions based on the emotional stress state.

Kappa statistics were used to assess inter-rater variability and agreement between the reviewers. A Kappa score of overall agreement of 0.72% was found, which provides a substantial agreement between the raters.

ELIGIBILITY:
Inclusion Criteria:

* All emergency call recordings involving OHCA in the capital region of Denmark in the time period 01.09.2018 - 01.11.2019

Exclusion Criteria:

* Emergency medical services (EMS)-witnessed OHCA
* Missing emergency call recording
* Caller not physically by patient's site

Age Groups: Child, Adult, Older Adult
Study Population: Bystander who call the emergency number in case of OHCA
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2022-03-10 (Estimated); Study Completion 2022-03-10 (Estimated)

PRIMARY OUTCOMES:
Time to first compression | 0-15 minutes
  Time from the emergency call starts to first chest compression

SECONDARY OUTCOMES:
Time to to recognition of cardiac arrest | 0-15 minuts
  Time from the emergency call starts to recognition of cardiac arrest
Dispatcher encouraging when giving instructions | 0-15 minuts
  Was the medical dispatcher motivating and encouraging when giving instructions (Yes/No)
Dispatcher assertive or passive when giving instructions | 0-15 minuts
  Was the medical dispatcher assertive or passive when giving instructions (Yes/No)
Dispatcher instruct on depth and speed of compressions | 0-15 minuts
  Did the medical dispatcher instruct on depth and speed of compressions (Yes/No)

CONTACTS AND LOCATIONS:
Overall Officials: Gitte Linderoth, PhD, Principal Investigator — Copenhagen Emergency Medical Services; Fredrik Folke, PhD, Prof, Study Chair — Copenhagen Emergency Medical Services; Annette Ersbøll, PhD, Prof, Study Chair — National Institute of Public Health, University of Southern Denmark
Locations (1):
- Copenhagen Emergency Medical Services, Copenhagen, Ballerup, Denmark